CLINICAL TRIAL: NCT03714529
Title: Phase IIa Trial With PD-L1 IO103 Vaccination With Montanide in Patients With Basal Cell Carcinoma
Brief Title: A Study of IO103 in Montanide Adjuvant for Basal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, jeanette kaae, MD PhD, Herlev and Gentofte Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCC1801
Record Dates: First submitted 2018-09-27; First posted 2018-10-22 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): The vaccine consists of 500µl of 100µg PD-L1 peptide, dissolved in DMSO and PBS reconstituted with 500 µl Montanide ISA-51.
  Patients will be vaccinated Q2W for 10 weeks, and a further 12 weeks if a clinical response is measured.
  Interventions: Biological: PD-L1

INTERVENTIONS:
Biological: PD-L1 — IO103 is a anti-cancer therapy consisting of a synthetic PD-L1-derived peptide.
  Other Names: IO103

SUMMARY:
A single center, open-label, phase IIa, single arm, window of opportunity trial with IO103 and Montanide adjuvant in patients with surgically resectable BCC.

DETAILED DESCRIPTION:
10 patients with BCC will be vaccinated with a peptide derived from the immune checkpoint molecule PD-L1. Patients will be vaccinated once every 2 weeks (Q2W) for 10 weeks and then evaluated for a clinical response.

Patients with clinical response to vaccination will continue with one vaccination once every 4 weeks (Q4W) for 12 weeks and thus receive 9 vaccinations in total over the course of 22 weeks.

Patients with no effect of treatment after 6 vaccinations will be treated with standard of care (SOC).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. At least 1 histological verified superficial or nodular basal cell carcinoma on the body or limbs of bigger than 14 mm in the longest diameter
3. Willing to provide three 4 mm biopsies from the lesion/lesions
4. Not previously treated with a hedgehog pathway inhibitor
5. For women of childbearing potential: Agreement to use contraceptive methods with a failure rate of < 1 % per year during the treatment period and for at least 150 days after the treatment. Safe contraceptive methods for women are birth control pills, intrauterine device, contraceptive injection, contraceptive implant, contraceptive patch or contraceptive vaginal ring.
6. For men: Agreement to use contraceptive measures and agreement to refrain from donating sperm
7. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial in accordance with ICH-GCP and local legislation prior to admission to the trial
8. Sufficient bone marrow function, i.e.

   1. Leucocytes ≥ 1,5 x 109
   2. Granulocytes ≥ 1,0 x 109
   3. Thrombocytes ≥ 20 x 109

2. Creatinine < 2.5 upper normal limit, i.e. < 300 μmol/l 3. Sufficient liver function, i.e.

1. ALAT < 2.5 upper normal limit, i.e. ALAT <112 U/l
2. Bilirubin < 30 U/l

Exclusion Criteria:

1. The patient has a history of life-threatening or severe immune related adverse events on treatment with another immunotherapy and is considered to be at risk of not recovering
2. The patient has a history of severe clinical autoimmune disease
3. The patient has a history of pneumonitis, organ transplant, human immunodeficiency virus positive, active hepatitis B or hepatitis C
4. The patient has any condition that will interfere with patient compliance or safety (including but not limited to psychiatric or substance abuse disorders)
5. The patient is pregnant or breastfeeding
6. The patient has an active infection requiring systemic therapy
7. The patient has received a live virus vaccine within 30 days of planned start of therapy
8. Known side effects to Montanide ISA-51
9. Significant medical disorder according to investigator; e.g. severe asthma or chronic obstructive lung disease, dysregulated heart disease or dysregulated diabetes mellitus
10. Concurrent treatment with other experimental drugs
11. Any active autoimmune diseases e.g. autoimmune neutropenia, thrombocytopenia or hemolytic anemia, systemic lupus erythematosus, scleroderma, myasthenia gravis, autoimmune glomerulonephritis, autoimmune adrenal deficiency, autoimmune thyroiditis etc.
12. Severe allergy or anaphylactic reactions earlier in life.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Clinical response | All patients were evaluated 3 Month after last vaccination
  Evaluation and measurement of target BCC in cm2. Clinical response is evaluated as change in tumor size in mm.
Disease control rate | After 6 vaccinations with IO103 (10 weeks)
  Defined as change of the largest diameter of target BCC
Immune responses | After 6 vaccinations with IO103 (10 weeks)
  Immune responses in biopsies from basal cell carcinomas (BCC). Analyses which will include (but are not restricted to): Immunosign®CR/Pan Cancer Immune panel (gene expression level of multiple immune genes); Halioseek® CD8/PDL1(PDL1/CD8, CD8+ quantification by digital pathology, PDL1+ tumoral cells and Immune cells analysis by a pathologist); Immunoscore (CD3 and CD8 immune histochemistry (IHC) testing, scanning and image analysis); MHC Class I and II (IHC, scanning and image analysis)

SECONDARY OUTCOMES:
Immune responses in skin | After 6 vaccinations with IO103 (10 weeks)
  Immune responses in skin delayed type hypersensitivity (DTH). Skin-infiltrating lymphocytes (SKILs) are tested for specificity to the PD-L peptides as a sign of induction of a functional immune response
Incidence of treatment emergent adverse events (safety and tolerability) | From the time that the subject provides written informed consent and throughout the trial duration, until 30 days post last dose of trial treatment
  Events will be recorded and graded using CTCAE version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Inge Marie Svane, Prof, Study Director — Herlev and Gentofte Hospital
Locations (1):
- Herlev and Gentofte Hospital, Hellerup, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Munir Ahmad S, Martinenaite E, Hansen M, Junker N, Borch TH, Met O, Donia M, Svane IM, Andersen MH. PD-L1 peptide co-stimulation increases immunogenicity of a dendritic cell-based cancer vaccine. Oncoimmunology. 2016 Jul 1;5(8):e1202391. doi: 10.1080/2162402X.2016.1202391. eCollection 2016 Aug. PMID 27622072